CLINICAL TRIAL: NCT03530943
Title: Efficacy of College-Based, Animal-Assisted Stress-Prevention Programs on Human and Animal Participants
Brief Title: Pet Partners for Promotion of Academic Life Skills
Acronym: Pet PALS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Washington State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 126634-001
Record Dates: First submitted 2018-03-20; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Stress Prevention; Cortisol; Anxiety Disorders and Symptoms; Depression Disorders and Symptoms; Executive Functioning; Motivation and Learning; Momentary Emotion; Study Strategies; Perceived Stress; Animal Behavior; Animal Stress; Dyadic Interaction; Alpha-amylase
MeSH Terms: conditions — Anxiety Disorders; Behavior, Animal

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants remained unaware of their treatment allocation until after completing the baseline (pretest) assessments and the onset of their intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Academic Stress Management (Active Comparator): Students assigned to the Academic Stress Management (ASM) condition will attend a series of once weekly, one hour long workshops over four consecutive weeks during which time they will receive 100% exposure to various evidence-based academic stress management tools.
  Interventions: Behavioral: Academic Stress Management tools
- Human Animal Interaction Enhanced (Experimental): Students assigned to the Human Animal Interaction - Enhanced (HAI-E) condition will attend a series of once weekly, one hour long workshops over four consecutive weeks. This group receives 50% exposure to structured and unstructured animal assisted activities and 50% exposure to various evidence-based academic stress management tools.
  Interventions: Behavioral: Animal Assisted Activities; Behavioral: Academic Stress Management tools
- Human Animal Interaction only (Experimental): Students assigned to the Human Animal Interaction - only (HAI-O) condition will attend a series of once weekly, one hour long workshops over four consecutive weeks. This group will be receive 100% exposure to structured and semi-structured animal assisted activities.
  Interventions: Behavioral: Animal Assisted Activities

INTERVENTIONS:
Behavioral: Animal Assisted Activities — Students interact with canines in small group settings under the supervision of their handlers during structured and semi-structured activities designed to strengthen physiological, emotion and behavioral regulation
  Arms: Human Animal Interaction Enhanced; Human Animal Interaction only
Behavioral: Academic Stress Management tools — Evidence-based workshops focus on evidence-based content and activities designed to enhance academic stress management knowledge and skills, motivation and learning, adaptive sleep, and study and test-taking behavior through strengthening physiological, emotion and behavioral regulation
  Arms: Academic Stress Management; Human Animal Interaction Enhanced

SUMMARY:
The current study utilized a randomized controlled trial, conducted in a real-life setting, to determine whether, how, under which conditions, and for whom, infusing various levels of human-animal interaction (HAI) in a 4-week, university-based stress prevention program provides an effective approach to prevent negative ramifications of university students stress, promote student executive functioning and learning, while safeguarding animal welfare. This study will examine effects of sole exposure to evidence-based stress prevention content, hands-on HAI with registered PET Partner teams, or combinations thereof on students' moment-to-moment well-being and longer-term functioning in socioemotional, cognitive and physiological domains.This study will also develop a comprehensive coding system and measure the dynamic nature of behavior of participants, handlers and animals during university- based animal assisted activities, as well as the HAI environment. The data and analyses will then be utilized to inform the development of a quantitative measure to capture of the quality of human animal interaction in various settings to experimentally determine causal pathways underlying program effects on humans and animals.

ELIGIBILITY:
Inclusion Criteria:

* Current enrollment at the campus

Exclusion Criteria:

* Children under 18 years old
* Prior history of animal abuse
* Participation in an an academic stress management workshop within 6 months of study participation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Salivary Cortisol (Diurnal) | Diurnal salivary cortisol was measured three times: at baseline one week before the intervention; at post-test one week following the conclusion of the intervention (baseline+5 weeks); and at follow-up six weeks after the posttest (baseline+11 weeks).
  Participants provided three samples (wakeup, afternoon, bedtime) over two consecutive days for a total of six samples.
Change in Salivary Cortisol (Basal) | Salivary cortisol was measured immediately preceding the beginning of each of the four programming sessions
Change in Salivary Cortisol (Momentary Reactivity) | Salivary cortisol was measured two to three times each of the four programming sessions in response to various program activities.
Change in Momentary Emotion (Experience Sampling Method Questionnaire) | Momentary emotion was measured three times each of the four programming sessions, immediately before entering the program area, and two additional times 30 and 50 minutes after the program start following various 10 minute activities
Change in Learning and Study Strategies (Learning and Study Strategies Inventory) | Learning and study strategies were measured three times: at baseline one week before the intervention; at post-test one week following the conclusion of the intervention (baseline+5 weeks); at follow-up six weeks after the posttest (baseline+11 weeks).
Change in Depression (Beck Depression Inventory) | Depression was measured three times: at baseline one week before the intervention; at post-test one week following the conclusion of the intervention (baseline + 5 weeks); and at follow-up six weeks after the posttest (baseline + 11 weeks).
Change in Anxiety (Beck Anxiety Inventory) | Anxiety was measured three times: at baseline one week before the intervention; at post-test one week following the conclusion of the intervention (baseline + 5 weeks); and at follow-up six weeks after the posttest (baseline + 11 weeks).
Change in Perceived Stress (Perceived Stress Scale - 10) | Perceived stress was measured three times: at baseline one week before the intervention; at post-test one week following the conclusion of the intervention (baseline + 5 weeks); and at follow-up six weeks after the posttest (baseline + 11 weeks).
  The Perceived Stress Scale -10 is a 10-item measure resulting in a single composite score ranging from 0 to 40 with higher scores representing higher levels of reported perceived stress.
Change in Executive Functioning (Behavior Rating Inventory of Executive Functioning - Adult Version) | Executive functioning was measured three times: at baseline one week before the intervention; at post-test one week following the conclusion of the intervention (baseline + 5 weeks); and at follow-up six weeks after the posttest (baseline + 11 weeks).

SECONDARY OUTCOMES:
Salivary Alpha-Amylase (Diurnal) | Diurnal salivary alpha-amylase was measured three times: at baseline one week before the intervention; at post-test one week following the conclusion of the intervention (baseline+5 weeks); and at followup six weeks after the posttest (baseline+11 weeks)
  Participants provided three samples (wakeup, afternoon, bedtime) over two consecutive days for a total of six samples.
Salivary Alpha-Amylase (Basal) | Salivary alpha-amylase was measured immediately preceding the beginning of each of the four programming sessions
Salivary Alpha-Amylase (Momentary Reactivity) | Salivary alpha-amylase was measured two to three times during each of the four programming sessions in response to various program activities.
Attitudes Towards Learning | Attitudes towards learning were measured three times: at baseline one week before the intervention; at post-test one week following the conclusion of the intervention (baseline+5 weeks); and at follow-up six weeks after the posttest (baseline+11 weeks)
Self-perceived worry (Penn State Worry Questionnaire) | Self-perceived worry was measured three times: at baseline one week before the intervention; at post-test one week following the conclusion of the intervention (baseline + 5 weeks); and at follow-up six weeks after the posttest (baseline + 11 weeks).

OTHER OUTCOMES:
Video observation coding | Recordings captured each dog-handler station, capturing 70-80 minutes throughout the program beginning 10 minutes before participants entry in the room through the end of each session.
  Video recordings capturing student, dog, and handler behaviors during the human-animal interaction sessions

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Pendry, PhD, Principal Investigator — Washington State University
Locations (1):
- Washington State University, Pullman, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pendry P, Carr AM, Gee NR, Vandagriff JL. Randomized Trial Examining Effects of Animal Assisted Intervention and Stress Related Symptoms on College Students' Learning and Study Skills. Int J Environ Res Public Health. 2020 Mar 15;17(6):1909. doi: 10.3390/ijerph17061909. PMID 32183453
- [Derived] Pendry P, Kuzara S, Gee NR. Evaluation of Undergraduate Students' Responsiveness to a 4-Week University-Based Animal-Assisted Stress Prevention Program. Int J Environ Res Public Health. 2019 Sep 10;16(18):3331. doi: 10.3390/ijerph16183331. PMID 31509993